CLINICAL TRIAL: NCT05314491
Title: A Prospective, Post-marketing Study Evaluating Clinical and Radiographic Early Outcomes of Total Knee Arthroplasty With Multigen Plus CCK Alone or Involving the AMF TT Cones.
Brief Title: Multigen Plus CCK and AMF TT Cones Follow Up Study
Status: Recruiting | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: K-24
Record Dates: First submitted 2022-03-30; First posted 2022-04-06 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Total Knee Arthroplasty; Revision Total Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Multigen Plus CCK
  Interventions: Device: Multigen Plus CCK
- Multigen Plus CCK in combination with AMF TT cones
  Interventions: Device: Multigen Plus CCK; Device: AMF TT cones

INTERVENTIONS:
Device: Multigen Plus CCK — Total Knee Arthroplasty
Device: AMF TT cones — To fill a proximal tibia or distal femur defect
  Groups: Multigen Plus CCK in combination with AMF TT cones

SUMMARY:
This study is aimed to provide a clinical and radiographic evaluation of 68 condylar-constrained Total Knee Arthroplasty (TKA) using a single type of prosthesis (Multigen Plus CCK configuration), alone or involving the AMF TT cones, in patients with joint instability or inadequate ligament function, both in complex primary and revision procedures.

DETAILED DESCRIPTION:
This is a post-market, multicentric, prospective, open label study. It is a post-marketing clinical study because the investigational devices are registered, CE marked, and used according to the intended use.

The assignment of any subject involved in the study is determined preoperatively by the aetiology evaluated by the Investigator and falls within the current practice. The decision to use this specific prosthesis design is decided by the Investigators independently and clearly separated from the decision to include the subject in the study.

Baseline measurements (pre-operative clinical assessment and radiographic analysis at discharge) serves as internal control for the assessment of post-operative data.

The study will be carried out in 3 sites in Europe for a total number of 68 study subjects, in whom the decision to implant the Multigen Plus CCK system, alone or in combination with the AMF TT cones, has been taken prior to, and independently from, the decision to include the subject in the study.

The enrolment is competitive until the required recruitment target is met.

The expected number of visits for each study subject is 6, and includes:

* a pre-operative visit (before the subject receives the Multigen Plus CCK system alone or involving the AMF TT cones).
* the intra-operative visit (that is the same day of the surgery).
* the discharge visit (after the surgery according to the clinical practice).
* the following follow-up visits: at 3 months, 12 months, and 24 months after the surgery.

All eligible subjects who agree to participate in the study will be recruited and monitored throughout the duration of the study. For each visit and for each single study subject, radiographic and clinical data will be assessed up to the 24-month follow-up visit according to the standard of care of the site, when applicable. Also, Adverse Events and Serious Adverse Events will be collected and assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age ≥ 18 years old.
* Given written informed consent approved by the reference Ethics Committee (EC).
* Subjects in whom a decision has already been made to perform a Total Knee Arthroplasty with Multigen Plus system as per Indication For Use. The decision to implant a Multigen Plus CCK system, alone or involving the AMF TT cones, must be taken prior to, and independently from, the decision to enrol the subject. This decision should be made in accordance with routine clinical practice at the study site concerned.
* Subjects able to comply with the Study Protocol.

Exclusion Criteria:

* Age < 18 years old.
* Subjects with any Multigen Plus system contraindication for use, or any AMF TT cones contraindication for use when used in combination with the Multigen Plus CCK, as reported in the current Instruction For Use.
* Any clinically significant pathology based on the medical history that the Investigator feels may affect the study evaluation.
* Female subjects who are pregnant, nursing, or planning a pregnancy.
* Previous knee replacement on the contralateral side within the last year and whose outcome is achieving an KSS < 70 points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population for this study includes adult subjects in whom the decision to perform a Total Knee Arthroplasty with Multigen Plus CCK system, alone or involving the AMF TT cones, must be taken prior to, and independently from, the decision to include the subject into the study.
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score (KSS) | Month 24
  Functional changes in the Knee Society Score (KSS) from pre-operative (baseline) to 2 years after the surgery.

SECONDARY OUTCOMES:
KOOS-ADL (Function in Daily Living subdomain) | Month 24
  Functional changes in the KOOS-ADL (Function in Daily Living subdomain) at 2 years after the surgery.
VISUAL ANALOGUE SCALE (VAS) PAIN | Month 24
  Changes in the VAS Pain score from pre-operative (baseline) to 2 years after the surgery. Scale is from 0 to 10, where 0 means NO PAIN and 10 VERY SEVERE PAIN.
Kaplan-Meier analysis | Month 24
  Survival rate of the implant (Kaplan-Meier estimate) at 2 years after the surgery.
Radiographic assessment | Month 24
  Radiographic implant evaluation and stability assessment at 2 years after the surgery.
Safety evaluation | Intra-operatively, Month 3, Month 12, and Month 24
  Incidence, type, and severity of all the Device Deficiency (DD), Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Device Effects (ADEs), and Serious Adverse Device Effects (SADEs) occurred at each follow-up

CONTACTS AND LOCATIONS:
Locations (3):
- Hospital Senhora da Oliveira in Guimarães, Guimarães, Portugal
- Saints Cyril and Methodius Hospital, Bratislava, Slovakia
- Royal Devon and Exeter Hospital, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No